CLINICAL TRIAL: NCT03910088
Title: Oral Pregabalin Versus Intravenous Hydrocortisone in Treatment of Postdural Puncture Headache After Spinal Anesthesia for Elective Cesarean Section
Brief Title: Pregabalin Versus Hydrocortisone for Postdural Puncture Headache After Spinal for Cesarean
Acronym: PDPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesrine El-Refai, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CairoU11112017
Record Dates: First submitted 2019-04-02; First posted 2019-04-10 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Post-Dural Puncture Headache
Keywords: spinal; cesarean; pregabalin
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Pregabalin; Capsules; Hydrocortisone; Acetaminophen; Fluid Therapy; Caffeine; Diclofenac

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): received conventional treatment in the form of good oral hydration, 500 mg of acetaminophen plus 65 mg of caffeine oral tablets thrice daily, 3 cups of coffee daily, 50 mg of diclofenac potassium oral tablets twice daily and recumbent positioning for 48 hours
  Interventions: Drug: Acetaminophen; Other: oral fluids; Drug: Caffeine; Drug: Diclofenac
- Pregabalin (Active Comparator): received the conventional treatment plus 100 mg of pregabalin oral tablet every 8 hours for 48 hours
  Interventions: Drug: Pregabalin 100Mg Oral Cap; Drug: Acetaminophen; Other: oral fluids; Drug: Caffeine; Drug: Diclofenac
- Hydrocortisone (Active Comparator): received the conventional treatment plus 100 mg of hydrocortisone IV every 8 hours for 48 hours.
  Interventions: Drug: Hydrocortisone; Drug: Acetaminophen; Other: oral fluids; Drug: Caffeine; Drug: Diclofenac

INTERVENTIONS:
Drug: Pregabalin 100Mg Oral Cap — giving a drug to relieve post-dural puncture headache
  Arms: Pregabalin
Drug: Hydrocortisone — Giving drug to relieve post-dural puncture headache
  Arms: Hydrocortisone
Drug: Acetaminophen — giving a drug to relieve post-dural puncture headache
  Other Names: Paracetamol
Other: oral fluids — giving oral fluids to maintain good hydration
  Other Names: good hydration
Drug: Caffeine — giving a drug to relieve post-dural puncture headache
Drug: Diclofenac — giving a drug to relieve post-dural puncture headache

SUMMARY:
Postdural puncture headache (PDPH) is a common complication after spinal anesthesia. The role of pregabalin and hydrocortisone in the treatment of PDPH is unclear. The aim of this work is to assess and compare the efficacy of both drugs in severe cases of PDPH after spinal anesthesia for elective cesarean section.

DETAILED DESCRIPTION:
The study will be done on 30 patient with PDPH with VAS score ≥ 5 after spinal anesthesia for elective cesarean section. Patients will be divided into three groups: Control group (group C):will receive conventional treatment in the form of good oral hydration, 500 mg of acetaminophen plus 65 mg of caffeine oral tablets thrice daily, 3 cups of coffee daily, 50 mg of diclofenac potassium oral tablets twice daily and recumbent positioning for 48 hours. Pregabalin group (group P): will receive the conventional treatment plus 100 mg of pregabalin oral tablet every 8 hours for 48 hours. Hydrocortisone group (group H): will receive the conventional treatment plus 100 mg of hydrocortisone IV every 8 hours for 48 hours. The three groups will be compared regarding the headache intensity using a visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective cesarean section under spinal anesthesia.
* Patients aged 18 to 40 years old.
* Patients classified as ASA I or II.

Exclusion Criteria:

* Patients with known sensitivity to any of the used drugs.
* Patients classified as ASA III or more.
* Preeclampsia.
* Patients with a history of chronic headache or migraine Patients receiving pregabalin for chronic pain.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study group is the pregnant females undergoing cesarean section
Enrollment: 30 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of pain using Visual Analogue Scale | the first 48 hours following treatment
  Headache intensity after 1 minute in upright position using the Visual Analogue Scale for pain assessment ranging from 0 to 10, with zero means no pain and 10 is the worst pain after 48 hours of treatment

SECONDARY OUTCOMES:
Assessment of the amount of rescue drug | The first 48 hours following treatment
  Total dose of nalbuphine given in each group..
incidence of side effects of the studied drug | the first 48 hours following treatment
  incidence of Somnolence
incidence of side effect of the studied drug | the first 48 hours following treatment
  incidence of dizziness

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Zamalek, Egypt

IPD SHARING:
Plan to Share IPD: No